CLINICAL TRIAL: NCT04667481
Title: Investigating Various Adaptive-Training Exercise Programs for Improving Cardiorespiratory Fitness After Breast Cancer Treatment (ACTIVATE)
Brief Title: Adaptive Training Exercise Programs for Improving Cardiorespiratory Fitness After Breast Cancer Treatment, The ACTIVATE Trial
Acronym: ACTIVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kerryn Reding, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1121129; P30CA015704 (NIH); 10872 (Other: Fred Hutch/University of Washington Cancer Consortium); NCI-2021-01114 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-11-09; First posted 2020-12-14 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Invasive Breast Carcinoma
Keywords: breast cancer; exercise; fatigue; fitness; aerobic; survivor
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (aerobic exercise) (Experimental): Patients participate in AE sessions 3 times per week for 12 weeks. After 12-weeks, non-responders participate in combined AE and RE sessions for an additional 12 weeks, while responders continue participating in the AE sessions alone for an additional 12 weeks.
  Interventions: Other: Aerobic Exercise Intervention; Other: Resistance Exercise Intervention; Other: Quality-of-Life Assessment
- Arm II (resistance exercise) (Experimental): Patients participate in RE sessions 3 times per week for 12 weeks. After 12-weeks, non-responders may participate in a further 12-weeks of combined AE and RE sessions, while responders continue participating in the RE sessions alone for an additional 12 weeks.
  Interventions: Other: Aerobic Exercise Intervention; Other: Resistance Exercise Intervention; Other: Questionnaire Administration; Other: Quality-of-Life Assessment
- Control Group (digital exercise interventions) (Experimental): After 24 weeks, patients receive a digital copy of the 12-week AE sessions and 12-week RE sessions and an outline of sessions for 24 weeks.
  Interventions: Other: Exercise Intervention: Digital copies and outline of sessions; Other: Questionnaire Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Aerobic Exercise Intervention — Participate in aerobic exercise intervention
  Arms: Arm I (aerobic exercise); Arm II (resistance exercise)
Other: Resistance Exercise Intervention — Participate in resistance exercise intervention
  Arms: Arm I (aerobic exercise); Arm II (resistance exercise)
Other: Exercise Intervention: Digital copies and outline of sessions — Receive digital copy of AE and RE sessions and an outline of sessions
  Arms: Control Group (digital exercise interventions)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm II (resistance exercise); Control Group (digital exercise interventions)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This clinical trial studies the feasibility of implementing various adaptive training exercise programs to improve cardiorespiratory fitness in patients after receiving breast cancer treatment. Information from this study may help researchers better understand how to implement adaptive training interventions to improve cardiorespiratory fitness in patients after receiving breast cancer treatment.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to the interventional groups or control group.

INTERVENTION GROUPS: Patients are randomized to 1 of 2 interventional arms.

ARM I: Patients participate in aerobic exercise (AE) sessions 3 times per week for 12 weeks. After 12-weeks, non-responders participate in combined AE and resistance exercise (RE) sessions for an additional 12 weeks, while responders continue participating in the AE sessions alone for an additional 12 weeks.

ARM II: Patients participate in RE sessions 3 times per week for 12 weeks. After 12-weeks, non-responders may participate in a further 12-weeks of combined AE and RE sessions, while responders continue participating in the RE sessions alone for an additional 12 weeks.

CONTROL GROUP: After 24 weeks, patients receive a digital copy of the 12-week AE sessions and 12-week RE sessions and an outline of sessions for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years, inclusive
2. Female gender
3. Prior diagnosis of invasive breast cancer
4. Completion of chemotherapy or receipt of trastuzumab (Herceptin) therapy within the past 6 - 60 months (0.5 - 5 years)
5. Reduced cardiorespiratory functional capacity, defined as below the median estimated CRF for age/sex-matched controls

Exclusion Criteria:

1. Actively receiving radiation treatment
2. Medical history of heart failure, coronary artery disease or arrhythmia
3. Contraindications to cardiopulmonary exercise testing (CPET)
4. Contraindications to magnetic resonance imaging (MRI) (e.g ferromagnetic cerebral aneurysm clips or other intraorbital/intracranial metal; pacemakers, defibrillators, functioning neurostimulator devices, non-compatible MRI tissue expanders or breast implants, or other implanted non-compatible MRI devices), weight over 550 lbs, or symptomatic claustrophobia
5. Contraindications to exercise, including a history of surgery with sequelae that restrict ability to exercise safely or comfortably
6. Unwilling to complete intervention procedures or outcome measures

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerryn W Reding, PhD, MPH, RN, Principal Investigator — University of Washington
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Resistance Exercise) | Control Group (Digital Exercise Interventions)
Started | 9 | 9 | 9
Completed | 9 | 8 | 8
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Resistance Exercise) | Control Group (Digital Exercise Interventions) | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 6 | 23
  >=65 years | 1 | 0 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (5.7) | 48.9 (11.7) | 56.6 (11.6) | 54.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 9 | 27
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 9 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 6 | 6 | 8 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility
Description: Will be determined with all-cause intervention discontinuation rate, which is the proportion of all intervention participants who permanently stop the intervention prior to week 24 for any reason.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Groups:
- Arm I: Aerobic Exercise: ARM I: Patients participate in aerobic exercise (AE) sessions 3 times per week for 12 weeks. After 12-weeks, non-responders participate in combined AE and resistance exercise (RE) sessions for an additional 12 weeks, while responders continue participating in the AE sessions alone for an additional 12 weeks.
- Arm II: Resistance Exercise: ARM II: Patients participate in RE sessions 3 times per week for 12 weeks. After 12-weeks, non-responders may participate in a further 12-weeks of combined AE and RE sessions, while responders continue participating in the RE sessions alone for an additional 12 weeks.
Arm/Group | Arm I: Aerobic Exercise | Arm II: Resistance Exercise
Number analyzed (Participants) | 9 | 9
Participants
  Discontinued Intervention | 1 | 3
  Completed Intervention | 8 | 6

2. Secondary Outcome: Intervention Safety: Adverse Events
Description: Intervention safety will be determined by reviewing and quantifying the number of adverse events (mild, moderate, or severe), serious adverse events, and by reviewing the type and severity of adverse events attributed to study procedures among each study group.
Time Frame: Up to 24 weeks
Population: Only adverse events probably or definitely attributed to study procedures are counted.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: Aerobic Exercise: ARM I: Patients participate in aerobic exercise (AE) sessions 3 times per week for 12 weeks. After 12-weeks, non-responders participate in combined AE and resistance exercise (RE) sessions for an additional 12 weeks, while responders continue participating in the AE sessions alone for an additional 12 weeks.
- Control Group: After 24 weeks, patients receive a digital copy of the 12-week AE sessions and 12-week RE sessions and an outline of sessions for 24 weeks.
  Exercise Intervention: Digital copies and outline of sessions: Receive digital copy of AE and RE sessions and an outline of sessions
  Questionnaire Administration: Ancillary studies
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Arm 1: Aerobic Exercise | Arm II: Resistance Exercise | Control Group
Number analyzed (Participants) | 9 | 9 | 9
Participants
  Count of participants with at least one AE | 2 | 3 | 0
  Gastrointestinal/Digestive | 0 | 0 | 0
  Respiratory | 0 | 1 | 0
  Skin | 0 | 0 | 0
  Musculoskeletal | 2 | 3 | 0
  Nervous System/Neurological | 0 | 0 | 0
  Psychiatric | 0 | 0 | 0
  Injuries | 1 | 2 | 0

3. Secondary Outcome: Study Feasibility
Description: Study feasibility will be measured by calculating recruitment rates (proportion of enrolled participants to all individuals approached), and loss to follow-up (proportion of participants who do not complete post-intervention assessments). A benchmark to determine feasibility is < 40% loss to follow-up.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- All Participants: Includes all participants randomized to either intervention or control
Arm/Group | All Participants
Number analyzed (Participants) | 27
Participants
  Did not complete endpoint assessment | 2
  Completed endpoint assessment | 25

4. Secondary Outcome: Intervention Acceptability
Description: Acceptability will be measured with qualitative, open-ended to assess participant experience in the intervention and gather information for improving the protocol in future studies. Of particular attention will be the tolerability of a remote, home-based exercise intervention with a semi supervised format.
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Aerobic Exercise | Arm II: Resistance Exercise
Number analyzed (Participants) | 9 | 9
Participants
  Satisfied with sessions | 9 | 9
  Exercise Provided Enough Challenge | 9 | 9
  Desired more personalized instruction | 3 | 4

5. Secondary Outcome: Intervention Session Intensity
Description: The Rating of Perceived Exertion (RPE) scale asks respondents to rate the intensity of exercise on a 1-10 scale, with higher values representing greater perceived exertion (1 = Very Light Activity, 10 = Maximum Possible Exertion). The measure has been validated for estimating both aerobic and resistance exercise exertion levels, providing a standard measure across intervention modalities. The average RPE for full-intensity sessions (the first few weeks involve an increasing RPE across sessions) will be calculated for each participant.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Resistance Exercise)
Number analyzed (Participants) | 9 | 9
units on a scale | 5.86 (1.37) | 5.60 (1.62)

6. Secondary Outcome: Intervention Adherence
Description: Participants will complete an RPE rating after each session. These ratings will be used to calculate adherence rate for each participant. A session with an RPE that is at or above the intended RPE will be considered adherent. The number of adherent sessions will be divided by the total number of sessions, whether the session was attended or not. The participant adherence rates will be averaged to find a mean adherence rate per participant.
Time Frame: Up to 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of adherent sessions
Arm/Group | Arm I (Aerobic Exercise) | Arm II (Resistance Exercise)
Number analyzed (Participants) | 9 | 9
percentage of adherent sessions | 52.8 (31.0) | 40.7 (32.2)

7. Other Pre Specified Outcome: Maximal Exercise Capacity (Absolute)
Description: This is operationalized as maximal exercise capacity, which is ascertained by measuring peak oxygen consumption (volume oxygen [VO2] peak) during cardiopulmonary exercise testing (CPET). All CPETs will be administered by a trained exercise physiologist using the Modified Bruce protocol, an appropriate testing paradigm for people with reduced physical functioning. This procedure will estimate the VO2 (absolute).
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Maximal Exercise Capacity (Relative to Bodyweight)
Description: This is operationalized as maximal exercise capacity, which is ascertained by measuring peak oxygen consumption (volume oxygen [VO2] peak) during cardiopulmonary exercise testing (CPET). All CPETs will be administered by a trained exercise physiologist using the Modified Bruce protocol, an appropriate testing paradigm for people with reduced physical functioning. This procedure will estimate the VO2 (relative to bodyweight).
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Submaximal Exercise Capacity
Description: Submaximal exercise capacity, also considered functional capacity, will be determined with the six minute walk test (6MWT), which measures the distance a person can walk in six minutes (6MWD). A widely used measure of submaximal exercise capacity, the 6MWT will be administered at all study timepoints to evaluate intervention response.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Anthropometrics (Weight)
Description: Prior to the measurement of body weight, participants will be instructed to remove heavy clothing and empty pockets of their contents. Weight will be measured to the nearest one-tenth kg with a calibrated balance beam or digital scale.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Anthropometrics (Hip Circumference)
Description: Hip circumference will be measured to the nearest one-tenth cm.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Anthropometrics (Height)
Description: Height will be measured while the participant stands without shoes using a wall-mounted stadiometer to the nearest one-tenth cm.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Abdominal Deposits of Fat
Description: Subcutaneous (SQ) fat and visceral adipose tissue (VAT) will be assessed via abdominal MRI. For analysis, fat depots will be separated into abdominal SQ fat and VAT which will be further segmented into intraperitoneal (IP) and retroperitoneal (RP) fat using commercially available software. SQ fat will be defined as the fat outside the muscular abdominal wall; IP fat as fat within the mesentery and omentum bounded anteriorly and laterally by the abdominal wall and posteriorly by a curved line drawn between the kidneys; RP fat as the remaining fat. Adipose tissues will be segmented and colored from other tissues based on pixel intensity and known divisions of tissue planes. The MRI analyst, blinded to participant characteristics, will correct any misidentified fat or non-fat regions using manual tools provided within the software. To calculate each of the compartmental fat deposits, the number of subpixels within each fat compartment.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Intermuscular Fat (IMF)
Description: The ratio of thigh IMF to skeletal muscle (SM) will be ascertained via magnetic resonance imaging (MRI) by trained MRI technologists. Participants will undergo a screening process with the MRI technologist to ensure that eligibility criteria for MRI scans are met. Participants will then change into a hospital gown and enter the MRI scanner. In this longitudinal assessment of IMF, the MRI technologist will be instructed to match participant scan positions across time by matching the current scan position with the participant's previous scan position, recorded at the timepoint prior. MRI analysts will quantitate total and compartment amounts of muscle and adipose tissue using cross-sectional areas of thigh skeletal muscle (SM) and IMF using commercially available software. Thigh IMF area will be calculated as the number of fat pixels within the thigh musculature multiplied by the pixel surface area.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Anthropometrics (Waist Circumference)
Description: Waist circumference will be measured to the nearest one-tenth cm.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change in Quality of Life
Description: The Short Form Health Survey-36 (SF-36) is a widely used self-report measure of quality of life and health status. Comprised of 36 multiple choice questions, the SF-36 queries general perceptions a participant has about their health, as well as limitations to physical activity, physical health problems, mental health problems, pain, and energy/fatigue. The SF-36 is used across health research domains, and in breast cancer has been validated as a reliable longitudinal monitor of quality of life.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Physical Activity and Sedentary Behaviors (IPAQ)
Description: Time spent engaging in physical activity will be measured with the Physical Activity Recall Interview. The PAR assesses time spent in physical activity over the past 7 days.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Perceived Well-being
Description: Participants' perception of their current well-being will be assessed with the 28-item 5-point Likert scale Functional Assessment of Cancer Therapy (FACT)-General. The FACT-G contains 4 subscales measuring physical, social, emotional, and functional well-being and has been validated for reliably measuring well-being in cancer patients.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Physical Activity and Sedentary Behaviors (SBQ)
Description: Time spent engaging in sedentary lifestyle behaviors will be measured with the self-administered Sedentary Behaviors Questionnaire (SBQ). The SBQ measures the minutes spent participating in 9 different sedentary behaviors per "typical" weekday and weekend day.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Level of Fatigue
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue scale is a 13-item scale originally developed for and widely used to assess cancer-related fatigue. The FACIT-Fatigue scale measures severity (i.e., "I feel fatigued"; "I feel weak all over") and impact of fatigue (e.g., "I need help doing my usual activities"; "I have to limit my social activity because I am tired") over the past week, with responses scored on a 5-point scale, from 0 "not at all" to 4 "very much." The FACIT-Fatigue scale has excellent psychometric properties and a focus on physical aspects of fatigue.
Time Frame: Up to 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected every 2 weeks for all 24 weeks of the intervention.
Description: Every two weeks, all participants were emailed a self-report survey to indicate the presence, severity, interference, and attribution of various medical symptoms
Arm/Group | Arm I: Aerobic Exercise | Arm II: Resistance Exercise | Control Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Aerobic Exercise (N=9) | Arm II: Resistance Exercise (N=9) | Control Group (N=9)
Any Gastrointestinal/Digestive (Gastrointestinal disorders) | 7 | 6 | 7
Any Skin (Skin and subcutaneous tissue disorders) | 5 | 5 | 5
Any Respiratory (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 3
Any Musculoskeletal (Musculoskeletal and connective tissue disorders) | 9 | 8 | 8
Any Neurological (Nervous system disorders) | 9 | 9 | 7
Any Psychiatric (Psychiatric disorders) | 6 | 5 | 6
Injury (Musculoskeletal and connective tissue disorders) | 7 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT04667481/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT04667481/ICF_000.pdf